CLINICAL TRIAL: NCT02883660
Title: Genecept Assay and Adverse Effects of Antidepressants
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 13P.25
Record Dates: First submitted 2016-02-24; First posted 2016-08-30 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Depression; Adverse Effects
Keywords: genetics; Antidepressants
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: patients who had empirically defined "increased AEs" on one of the specified antidepressants (SSRIs/ SNRIs). This group will get the Genecept Assay, which is a battery of pharmacogenetic tests relevant to psychiatry.
  Interventions: Genetic: Genocept Assay
- Controls: patients who did not have empirically defined "increased AEs" with an index antidepressant (one of the specified SSRIs/ SNRIs) AND were "nonresponders" to that antidepressant. This group will get the Genecept Assay, which is a battery of pharmacogenetic tests relevant to psychiatry.
  Interventions: Genetic: Genocept Assay

INTERVENTIONS:
Genetic: Genocept Assay — battery of pharmacogenetic tests relevant to psychiatry

SUMMARY:
The purpose of this study is to determine whether patients who have been prescribed antidepressant medications and have experienced significant adverse effects are more likely to be poor metabolizers on the CYP450 (CYP2B6, CYP2D6, CYP2C19, CYP3A4/5+) drug metabolizing enzymes and/or homozygous for the short allele of the serotonin transporter (SLC6A4) compared to patients who took an antidepressant medication and did not experience significant adverse effects but also had minimal or no response to the medication. The target medications being studied include escitalopram, citalopram, paroxetine, fluvoxamine, venlafaxine, duloxetine, bupropion, vortioxetine, vilazodone, and levomilnacipran only.

DETAILED DESCRIPTION:
Genetic variations in the CYP2B6, CYP2D6, CYP2C19, and CYP3A4/5+ drug metabolizing enzymes are responsible for metabolism of a large number of psychiatric and nonpsychiatric medications. Variations in the genes encoding for these enzymes can alter their activity resulting in unexpectedly high or low serum levels of the drug leading potentially to change in both efficacy and adverse events. The serotonin transporter protein is a presynaptic transmembrane protein responsible for serotonin reuptake. The "short" form of the serotonin transporter promoter (SLC6A4) is associated with reduced activity of the of the transporter. Patients who are homozygous for the "short" alleles of SLC6A4 may be more likely to have with poor response, slow response, and greater adverse events with serotonergic medications. The target medications being studied include escitalopram, citalopram, paroxetine, fluvoxamine, venlafaxine, duloxetine, bupropion, vortioxetine, vilazodone, and levomilnacipran only.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to give informed consent prior to the initiation of any protocol required procedures.
3. Subject must be able to understand the nature of the study, agree to comply with the study procedures, and communicate about medical history to the study personnel.
4. Subject was treated with one of the following "target antidepressants:" Escitalopram, citalopram, paroxetine, fluvoxamine, venlafaxine, duloxetine, bupropion, vortioxetine, vilazodone, and levomilnacipran. Rationale: These antidepressants are primarily metabolized by CYP isoenzymes that will be assessed. Antidepressants like sertraline, fluoxetine, and mirtazapine are metabolized by multiple CYP isoenzymes and therefore are less likely to be significantly affected by metabolizer status on a particular CYP isoenzyme. For patients who have been treated with multiple antidepressants, the antidepressant that was associated with the greatest overall burden of AEs will be selected as the target antidepressant.

5a. Study group: "Increased AEs" currently or in the past on one of the target antidepressants as operationally defined as either A or B: A) One or more AEs that were moderate/severe OR three or more AEs that were mild occurring on less than the usual minimum recommended dose of the antidepressant, or B) Three or more AEs that were moderate/severe OR five or more AEs that were mild on a dose of the antidepressant within the usual recommended dose 5b. Control group: Both A and B A. Less than 30% reduction in the severity of depression after treatment for at least 6 weeks B. Minimal or no AEs on that antidepressant

Exclusion Criteria:

1. Subjects on antidepressants other than those specified in the inclusion criteria.
2. Subjects for whom it is unclear which medication caused the adverse events
3. Subjects for whom participation in the study would be detrimental to their mental of physical health based on investigator's opinion
4. Subjects who have had a medical condition that, in the investigator's judgment, may be causing the reported adverse events
5. Prisoners or patients who are involuntarily incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred (100) subjects aged 18 years or older, currently or in the past on one of the target antidepressants, will be recruited into this study.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-02; Primary Completion 2017-07-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Poor metabolizers have more side effects | through study completion, approximately 2 years
  Our primary aim is to test the hypothesis that a statistically significantly higher proportion of Cases than Controls will be poor metabolizers on CYP450 isoenzymes (CYP2B6, CYP2D6, CYP2C19, CYP3A4/5+).
Homozygenous for short allele of SLC6A4 will result in more side effects | through study completion, approximately 2 years
  Our co-primary aim is to test the hypothesis that a statistically significantly higher proportion of Cases than Controls will be homozygenous for the short allele of SLC6A4.

CONTACTS AND LOCATIONS:
Overall Officials: William Jangro, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
no plan to make IPD available